CLINICAL TRIAL: NCT05479422
Title: European Clinical Registry for Optilume Urethral Drug Coated Balloon
Brief Title: Optilume Registry for Treatment of Stricture of the Anterior Urethra
Status: Active, not recruiting | Type: Observational
Sponsor: European Association of Urology Research Foundation (Other)
Collaborators: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR1276-001
Record Dates: First submitted 2022-06-27; First posted 2022-07-29 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Anterior Urethral Stricture, Male
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment of stricture of the anterior urethra with optilume DCB: Standard of care treatment of stricture of the anterior urethra using the Optilume Drug Coated Balloon.

SUMMARY:
The purpose of this registry is verifying the continued safety and effectiveness of the Optilume DCB clinical use in patients undergoing dilation of the urethral stricture.

DETAILED DESCRIPTION:
After being informed about the registry and potential risks, all patients providing written informed consent will undergo urethral dilation using the Optilume Drug Coated Balloon (standard of care procedure).

At 3, 6, 12 months, and annually 2 to 5 years after treatment patients will be invited to return to the hospital and several assessments will be performed, including questionnaires, if this is part of their standard care.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥ 18 years old
2. Subject diagnosed with a recurrent stricture ≤3cm in the anterior urethra that plans to be treated with Optilume® DCB in accordance with the approved Instructions for Use.
3. Subject provides written informed consent using an approved Informed Consent Form (ICF) and is willing to comply with standard follow-up assessments.

Exclusion Criteria:

1. Subjects with a known hypersensitivity to paclitaxel or structurally related compounds.
2. Subject is unwilling to abstain or use a condom for 30 days after the procedure.
3. Subject is unwilling to use highly effective contraception for 6 months after the procedure if partner is of childbearing potential.
4. Subjects with a history of carcinoma of the genitourinary system (e.g., kidney, bladder, prostate, urethra, testes) that is not considered in complete remission.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male subjects (≥ 18 years old) with a recurrent anterior urethral stricture
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2029-08-15 (Estimated); Study Completion 2029-08-15 (Estimated)

PRIMARY OUTCOMES:
Responder Rate at 12 Months | 12 months
  The responder rate is defined as the proportion of subjects experiencing a ≥30% improvement in International Prostate Symptom Score (IPSS) without repeat intervention for the study stricture. The responder rate at 12 months post-treatment will be compared against a performance goal of 60%.
  The International Prostate Symptom Score (IPSS) (score 0-7 = mild; score 8-19 = mediate; score 20-35 = severe complaints) was chosen as the primary patient-reported outcome measure (PROM) for follow-up due to its inclusion in the EAU guidelines, its long history of use, its inclusion as the primary PROM in the ROBUST clinical program, and the availability of literature describing clinically meaningful improvement in the setting of bladder outlet obstruction.
Rate of Treatment Related Serious Adverse Events at 3 months | 3 months
  The primary safety endpoint is defined as the proportion of subjects experiencing a treatment related Serious Adverse Event (SAE) through 3 months post-treatment. The primary safety endpoint will be analyzed with descriptive statistics and nominal 95% confidence interval.
  No single event type is expected to happen with greater frequency than other endoscopic therapies, therefore any event that meets the definition of an SAE and is considered treatment related will be included in the endpoint.

SECONDARY OUTCOMES:
Frequency and Severity of Treatment Related Adverse Events | Through study completion, an average of 3 years
  The proportion of subjects experiencing treatment related adverse events will be summarized by event type and severity as graded by the Clavien-Dindo scale. 'Treatment Related' consists of events deemed Possible, Probable, or Definite in relation to the Optilume® DCB or the dilation procedure.
Freedom from Repeat Intervention | Through study completion, an average of 3 years
  Defined as freedom from any reintervention for the stricture treated during the index procedure, including but not limited to:
  * Urethroplasty
  * Dilation with sounds, bougies, balloon, etc.
  * Direct vision internal urethrotomy
  * Dilation with the Optilume® DCB
  * Intermittent self-dilation / Clean Intermittent Catheterization (CIC)
  * Indwelling catheter (urethral or suprapubic)
  * Urethral stent
Anatomic Evaluation | Through study completion, an average of 3 years
  Outcomes related to anatomic recurrence of the stricture will be summarized via descriptive statistics. Anatomic recurrence will be defined as urethral lumen <14F measured by the inability to pass a flexible cystoscope or as measured via urethrogram. Outcomes will be reported as those free from stricture recurrence utilizing both definitions, as well as reported separately for those undergoing cystoscopy and those undergoing urethrography.

CONTACTS AND LOCATIONS:
Overall Officials: Nadir I. Osman, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (13):
- AZ Middelares, Ghent, Belgium
- Italy (3):
  - Department of Urology - San Raffaele University, Milan
  - AOU "Città della Salute e della Scienza" University of Turin, Torino
  - AOUI Verona, Urology Unit, Verona
- Oslo university hospital Rikshospitalet, Oslo, Norway
- Spain (3):
  - Marques de Valdecilla University Hospital, Santander, Cantabria
  - Lyx I Instituto de Urología, Madrid
  - Hospital Universitario de Navarra, Pamplona
- United Kingdom (5):
  - Epsom and St Helier Hospitals, Carshalton
  - Frimley Park Hospital, Frimley Health NHS Foundation Trust, Frimley
  - Freeman Hospital, Newcastle upon Tyne
  - Norfolk & Norwich University Hospital, Norwich
  - Sheffield Teaching Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No